CLINICAL TRIAL: NCT03818347
Title: Hydrogen Gas Immunotherapy Promotes the Rehabilitation and Prognosis of Cancer Patients After Standard Treatments
Brief Title: Hydrogen Gas for Cancer Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shanghai Asclepius Meditech Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Hydrogen-cancer
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-06

CONDITIONS: Adult Solid Tumor
Keywords: Solid tumor; Hydrogen gas

STUDY DESIGN:
Intervention Model Description: the patients will inhale hydrogen and oxygen with oxyhydrogen generator
Who Masked: Investigator
Masking Description: the experimental and control machines are of the same appearance and gas generation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxyhydrogen generator (AMS-H-03) (Experimental): Model: AMS-H-03 Rated gas output (L) : 3L/min, concentration of hydrogen and the oxygen was 66.6% and 33.3%, respectively In this group, the patients will inhale hydrogen and oxygen with oxyhydrogen generator. The check indexes are questionnaire of sleep, diet and exercise, CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Device: oxyhydrogen generator (AMS-H-03)
- Control (Placebo Comparator): In this group, the patients will inhale normal air with analogue machine. The check indexes are questionnaire of sleep, diet and exercise, CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Device: analogue machine

INTERVENTIONS:
Device: oxyhydrogen generator (AMS-H-03) — Rated gas output (L) : 3L/min, concentration of hydrogen and the oxygen was 66.6% and 33.3%, respectively. The patients inhale 3 hours each day through a cannula or mask, and persist for long term
  Other Names: hydrogen generator
  Arms: oxyhydrogen generator (AMS-H-03)
Device: analogue machine — This machine has the same apperance and gas condition
  Arms: Control

SUMMARY:
The aim of this study is the efficacy of hydrogen gas immunotherapy to rehabilitation and prognosis of cancer patients.

DETAILED DESCRIPTION:
By enrolling patients of multiple kinds of cancer adapted to enrolled criteria, this study will document for the first time the short and long term efficacy of hydrogen gas.The evaluation indexes include peripheral blood lymphocyte immunoassay, improvement of sleep, diet and exercise, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Standard therapies have finished according to NCCN guidelines or the patient refuses standard therapies
* Body tumor 1-6, the maximum tumor length < 2 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-02 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Improvement of sleep, diet and exercise | 3 months
  It will be evaluated by the questionnaire of EORTC QLQ-C30. The scores of each index before and after treatment need to be analyzed by statistical methods to reach a conclusion, and P< 0.05 is considered to be statistically different
Improvement of immune function | 3 months
  It will be evaluated by the blood test, including tumor marker alpha fetoprotein (AFP), lymphocyte subsets (T and NK cells) and circulating tumor cell (CTCs). The reference range of AFP is 0-40 IU/mL, higher than this range indicates tumor risk, and the higher the value is, the faster the tumor growth rate will be. The t-cell range of the lymphocyte subclass is 603-2990 cell/uL, and the NK cell range is 95-640 cell/uL, lower than the reference range indicates low immune function. The CTC reference range is 0-1, and higher than the reference range indicates tumor activity.

SECONDARY OUTCOMES:
Progress free survival（PFS） | 1 year
  follow-up of CT scan
Overall survival（OS） | 3 years
  follow-up survival

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Fuda cancer institute, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Chen JB, Kong XF, Qian W, Mu F, Lu TY, Lu YY, Xu KC. Two weeks of hydrogen inhalation can significantly reverse adaptive and innate immune system senescence patients with advanced non-small cell lung cancer: a self-controlled study. Med Gas Res. 2020 Oct-Dec;10(4):149-154. doi: 10.4103/2045-9912.304221. PMID 33380580
- [Derived] Chen JB, Kong XF, Mu F, Lu TY, Lu YY, Xu KC. Hydrogen therapy can be used to control tumor progression and alleviate the adverse events of medications in patients with advanced non-small cell lung cancer. Med Gas Res. 2020 Apr-Jun;10(2):75-80. doi: 10.4103/2045-9912.285560. PMID 32541132
- [Derived] Chen J, Kong X, Mu F, Lu T, Du D, Xu K. Hydrogen-oxygen therapy can alleviate radiotherapy-induced hearing loss in patients with nasopharyngeal cancer. Ann Palliat Med. 2019 Nov;8(5):746-751. doi: 10.21037/apm.2019.11.18. PMID 31865734